CLINICAL TRIAL: NCT02906202
Title: A Phase 3 Single Arm Study Evaluating the Efficacy and Safety of Gene Therapy in Subjects With Transfusion-dependent β-Thalassemia, Who do Not Have a β0/β0 Genotype, by Transplantation of Autologous CD34+ Stem Cells Transduced Ex Vivo With a Lentiviral βA-T87Q-Globin Vector in Subjects ≤50 Years of Age
Brief Title: A Study Evaluating the Efficacy and Safety of the LentiGlobin® BB305 Drug Product in Participants With Transfusion-Dependent β-Thalassemia, Who do Not Have a β0/β0 Genotype
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genetix Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGB-207
Record Dates: First submitted 2016-08-19; First posted 2016-09-20 (Estimated); Results first posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Beta-Thalassemia
MeSH Terms: conditions — beta-Thalassemia | interventions — betibeglogene autotemcel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LentiGlobin BB305 Drug Product (Experimental): Participants aged less than or equal to (<=) 50 years received a single intravenous (IV) infusion of LentiGlobin BB305 Drug Product at a dose of greater than or equal to (>=) 5.0*10^6 CD34 plus (+) cells per kilogram (cells/kg) following myeloablative conditioning with busulfan (termed the Transplant population).
  Interventions: Genetic: LentiGlobin BB305 Drug Product

INTERVENTIONS:
Genetic: LentiGlobin BB305 Drug Product — LentiGlobin BB305 Drug Product is administered by IV infusion following myeloablative conditioning with busulfan.
  Other Names: betibeglogene autotemcel

SUMMARY:
This is a single-arm, multi-site, single-dose, Phase 3 study in 23 participants less than or equal to (<=) 50 years of age with transfusion-dependent β-thalassemia (TDT), also known as β-thalassemia major, who do not have a β0 mutation at both alleles of the hemoglobin β (HBB) gene. The study will evaluate the efficacy and safety of autologous hematopoietic stem cell transplantation (HSCT) using LentiGlobin BB305 Drug Product.

ELIGIBILITY:
Inclusion Criteria:

* Participants <= 50 years of age at the time of consent or assent (as applicable), and able to provide written consent (adults, or legal guardians, as applicable) or assent (adolescents or children). Provided that the Data Monitoring Committee (DMC) has approved enrolling participants younger than 5 years of age, participants younger than 5 years of age may be enrolled if they weigh a minimum of 6 kilograms (kg) and are reasonably anticipated to be able to provide at least the minimum number of cells required to initiate the manufacturing process.
* Diagnosis of TDT with a history of at least 100 milliliter per kilogram per year (mL/kg/year) of pRBCs in the 2 years preceding enrollment (all participants), or be managed under standard thalassemia guidelines with >= 8 transfusions of pRBCs per year in the 2 years preceding enrollment (participants >= 12 years).
* Clinically stable and eligible to undergo (HSCT).
* Treated and followed for at least the past 2 years in a specialized center that maintained detailed medical records, including transfusion history.

Exclusion Criteria:

* Presence of a mutation characterized as β0 mutation at both alleles of the β-globin gene HBB.
* Positive for presence of human immunodeficiency virus type 1 or 2 (HIV-1 and HIV-2), hepatitis B virus (HBV), or hepatitis C (HCV).
* A white blood cell (WBC) count less than (<) 3×10^9/Liter (L), and/or platelet count < 100×10^9/L not related to hypersplenism.
* Uncorrected bleeding disorder.
* Any prior or current malignancy.
* Immediate family member with a known Familial Cancer Syndrome.
* Prior HSCT.
* Advanced liver disease.
* A cardiac T2* < 10 ms by MRI.
* Any other evidence of severe iron overload that, in the Investigator's opinion, warrants exclusion.
* Participation in another clinical study with an investigational drug within 30 days of Screening.
* Any other condition that would render the participant ineligible for HSCT, as determined by the attending transplant physician or investigator.
* Prior receipt of gene therapy.
* Pregnancy or breastfeeding in a postpartum female or absence of adequate contraception for fertile participant.
* A known and available Human leukocyte antigen (HLA) matched family donor.
* Any contraindications to the use of granulocyte colony stimulating factor (G-CSF) and plerixafor during the mobilization of hematopoietic stem cells and any contraindications to the use of busulfan and any other medicinal products required during the myeloablative conditioning, including hypersensitivity to the active substances or to any of the excipients.

Ages: 0 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2016-08-08 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Himal Lal Thakar, MD, Study Director — Genetix Biotherapeutics Inc.
Locations (8):
- United States (3):
  - Oakland, California
  - Chicago, Illinois
  - Philadelphia, Pennsylvania
- Marseille, France
- Hanover, Germany
- Rome, Italy
- Bangkok, Thailand
- London, United Kingdom

REFERENCES:
- [Derived] Locatelli F, Thompson AA, Kwiatkowski JL, Porter JB, Thrasher AJ, Hongeng S, Sauer MG, Thuret I, Lal A, Algeri M, Schneiderman J, Olson TS, Carpenter B, Amrolia PJ, Anurathapan U, Schambach A, Chabannon C, Schmidt M, Labik I, Elliot H, Guo R, Asmal M, Colvin RA, Walters MC. Betibeglogene Autotemcel Gene Therapy for Non-beta0/beta0 Genotype beta-Thalassemia. N Engl J Med. 2022 Feb 3;386(5):415-427. doi: 10.1056/NEJMoa2113206. Epub 2021 Dec 11. PMID 34891223
- [Derived] Hamed EM, Meabed MH, Aly UF, Hussein RRS. Recent Progress in Gene Therapy and Other Targeted Therapeutic Approaches for Beta Thalassemia. Curr Drug Targets. 2019;20(16):1603-1623. doi: 10.2174/1389450120666190726155733. PMID 31362654

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 9 centers from 08 August 2016 to 31 March 2022.
Pre-assignment Details: A total of 24 participants initiated mobilization procedure, of which 23 participants aged less than or equal to (<=) 50 years were treated with LentiGlobin BB305 Drug Product. As appropriate, data were analyzed at times based on Intent-to-Treat (ITT) population which included all 24 participants who initiated mobilization procedure.
Groups:
- LentiGlobin BB305 Drug Product: Participants aged <= 50 years received a single intravenous (IV) infusion of LentiGlobin BB305 Drug Product at a dose of greater than or equal to (>=) 5.0*10^6 CD34 plus (+) cells per kilogram (cells/kg) following myeloablative conditioning with busulfan (termed the Transplant population).
Period: Overall Study
Arm/Group | LentiGlobin BB305 Drug Product
Started | 24
Transplant Population | 23
Completed | 23
Not Completed | 1
Not completed — Discontinued after mobilization due to pregnancy | 1

BASELINE CHARACTERISTICS:
Population: ITT population included all participants who initiated mobilization procedure. As appropriate, data were analyzed at times based on ITT population which included all 24 participants who initiated any study procedures, beginning with mobilization by G-CSF and/or plerixafor.
Groups:
- LentiGlobin BB305 Drug Product: Participants aged <= 50 years received a single IV infusion of LentiGlobin BB305 Drug Product at a dose of >= 5.0*10^6 CD34+ cells/kg following myeloablative conditioning with busulfan (termed the Transplant population).
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: Years] | 15.0 [4 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Meet the Definition of Transfusion Independence (TI)
Description: TI was defined as a weighted average hemoglobin (Hb) >= 9 grams per deciliter (g/dL) without any packed red blood cell (pRBC) transfusions for a continuous period of >= 12 months at any time during the study after drug product infusion.
Time Frame: From 14 to 24 months post-transplant
Population: Transplant Population (TP) included all participants who received beti-cel. All participants in the TP (23 participants) were evaluable for TI.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 23
Percentage of participants | 91.3 [72.0 to 98.9]

2. Secondary Outcome: Percentage of Participants Who Meet the Definition of Transfusion Independence (TI) at Month 24
Description: TI was defined as a weighted average hemoglobin (Hb) >= 9 grams per deciliter (g/dL) without any packed red blood cell (pRBC) transfusions for a continuous period of >= 12 months at any time during the study after drug product infusion. Percentage of participants who met the definition of TI at Month 24 were evaluated
Time Frame: At Month 24 post-transplant
Population: TP included all participants who received beti-cel. All participants in the TP (23 participants) were evaluable for TI.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 23
Percentage of participants | 91.3 [72.0 to 98.9]

3. Secondary Outcome: Duration of Transfusion Independence (TI)
Description: Duration of TI was calculated as the time from the start of TI (that is (i.e.), first Hb >=9 with no transfusions in the preceding 60 days) up to the last available Hb at which the TI criteria are still met using Kaplan-Meier methodology. Duration of TI from start of TI up to Month 24 months was reported.
Time Frame: From start of TI up to Month 24
Population: TP included all participants who received beti-cel. All participants in the TP (23 participants) were evaluable for TI. Here, "Overall number of participants analyzed" signifies those participants who achieved TI (i.e. 21 participants as 2 participants did not achieve TI).
Measure: Median (Full Range); unit: months
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 21
months | 20.50 [18.2 to 22.5]

4. Secondary Outcome: Time From Drug Product Infusion to Achievement of Transfusion Independence (TI)
Description: Time from drug product infusion to achievement of TI was calculated as the time from drug product infusion to the first hemoglobin at which a participant can be declared as TI (that is to 'start of TI + >= 12 months', dependent on Hb lab schedule).
Time Frame: From 14 months post-drug product infusion through Month 24
Population: as for outcome 3
Measure: Median (Full Range); unit: months
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 21
months | 15.51 [14.8 to 19.4]

5. Secondary Outcome: Weighted Average Hemoglobin (Hb) During Transfusion Independence (TI)
Description: Weighted average Hb was defined as the weighted average of Hb values without any pRBC transfusions in the proceeding 60 days. The ratio of the time between two Hb values and the time between the first and the last Hb values was used as the weight for calculation.
Time Frame: From 60 days after the last pRBC transfusion through Month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 21
grams per deciliter (g/dL) | 11.473 (1.0395)

6. Secondary Outcome: Percentage of Participants Who Had a Reduction of At Least 50%, 60%, 75%, 90% or 100% in the Annualized pRBCs Transfusion Volume
Description: Percentage of participants reduction in the annualized mL/kg pRBCs transfused from 12 months post-drug product infusion through Month 24 (approximately a 12-month period) of at least 50%, 60%, 75%, 90% or 100% compared to the annualized mL/kg pRBC transfusion requirement during the 24 months prior to enrollment.
Time Frame: 12 months post-drug product infusion through Month 24
Population: TP included all participants who received beti-cel.
Measure: Number; unit: percentage of participants
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 23
percentage of participants
  Reduction at >= 50% | 95.7
  Reduction at >= 60% | 91.3
  Reduction at >= 75% | 91.3
  Reduction at >= 90% | 91.3
  Reduction at 100% | 91.3

7. Secondary Outcome: Annualized Number of pRBC Transfusions
Description: Annualized number of pRBC transfusions from 12 months post-drug product infusion through Month 24 were reported.
Time Frame: From 12 months post-drug product infusion through Month 24
Population: TP included all participants who received beti-cel.
Measure: Mean (Standard Deviation); unit: pRBC transfusions per year
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 23
pRBC transfusions per year | 0.95 (3.195)

8. Secondary Outcome: Annualized Volume of pRBC Transfusions
Description: Annualized volume of pRBC transfusions from 12 months post-drug product infusion through Month 24 was reported.
Time Frame: From 12 months post-drug product infusion through Month 24
Population: TP included all participants who received beti-cel.
Measure: Mean (Standard Deviation); unit: milliliter/kilogram/year (mL/kg/year)
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 23
milliliter/kilogram/year (mL/kg/year) | 11.607 (40.2964)

9. Secondary Outcome: Time From Drug Product Infusion to Last pRBC Transfusion
Description: Time from drug product infusion to last pRBC transfusion was reported.
Time Frame: From start of drug product infusion up to Month 24
Population: TP included all participants who received beti-cel.
Measure: Median (Full Range); unit: months
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 23
months | 0.953 [0.46 to 23.98]

10. Secondary Outcome: Time From Last pRBC Transfusion to Month 24
Description: Time From Last pRBC Transfusion to Month 24 was reported.
Time Frame: From last pRBC Transfusion up to Month 24 (actual maximum time frame of up to approximately 27 months due to visit window)
Population: TP included all participants who received beti-cel. Data are presented through the Month 24 Visit based on calendar dates and including visit windows. Notably due to institutional COVID-19 restrictions and scheduling conflicts one participant had a Month 24 visit 42 days out of this window.
Measure: Median (Full Range); unit: months
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 23
months | 23.228 [0.07 to 26.64]

11. Secondary Outcome: Weighted Average Nadir Hemoglobin (Hb)
Description: The weighted average nadir Hb was defined as the most recent Hb prior to each pRBC transfusion, on the day of transfusion or within 3 days and, if there was a period of more than 60 days without transfusion, all Hb records between Day 61 and last follow-up or next transfusion (inclusive) was included. The weighted average nadir Hb during the period of 12 months post-drug product infusion to Month 24 was compared to the weighted average nadir Hb during the 24 months prior to enrollment.
Time Frame: 12 months post-drug product infusion through Month 24
Population: TP included all participants who received beti-cel.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 23
g/dL | 9.546 (0.7007)

12. Secondary Outcome: Unsupported Total Hb Levels at Month 6, 9, 12, 18 and 24
Description: Unsupported total Hb level was defined as the total Hb measurement level without any acute or chronic pRBC transfusions within 60 days prior to the measurement date.
Time Frame: At Month 6, 9, 12, 18 and 24
Population: TP included all participants who received beti-cel. Here, "Overall number of participants analyzed" signifies those participants who had a least 1 unsupported total Hb measurement during Study HGB-207 and "number analyzed" signifies those participants who had an unsupported total Hb measurement at the specific timepoint.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 22
g/dL
  At Month 6 | 11.24 (1.249)
  At Month 9 | 11.22 (1.138)
  At Month 12: number analyzed (Participants) | 21
  At Month 12 | 11.45 (1.314)
  At Month 18: number analyzed (Participants) | 19
  At Month 18 | 11.80 (1.167)
  At Month 24: number analyzed (Participants) | 20
  At Month 24 | 11.77 (1.224)

13. Secondary Outcome: Number of Participants With Unsupported Total Hb Levels (>=10 g/dL, >=11 g/dL, >=12 g/dL, >=13 g/dL, and >=14 g/dL) at Months 6, 9, 12, 18 and 24
Description: The number of participants with unsupported total Hb levels (>=10 g/dL, >=11 g/dL, >=12 g/dL, >=13 g/dL, and >=14 g/dL) meeting the thresholds were reported at at Months 6, 9, 12, 18 and 24. Participants were evaluable if they had an unsupported total Hb measurement at the specific timepoint, where unsupported total Hb level is defined as the total Hb measurement level without any acute or chronic pRBC transfusions within 60 days prior to the measurement date.
Time Frame: At Month 6, 9, 12, 18 and 24
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 22
Participants
  At Month 6 (>=10 g/dL) | 17
  At Month 6 (>=11 g/dL) | 15
  At Month 6 (>=12 g/dL) | 7
  At Month 6 (>=13 g/dL) | 1
  At Month 6 (>=14 g/dL) | 0
  At Month 9 (>=10 g/dL) | 20
  At Month 9 (>=11 g/dL) | 14
  At Month 9 (>=12 g/dL) | 5
  At Month 9 (>=13 g/dL) | 1
  At Month 9 (>=14 g/dL) | 0
  At Month 12 (>=10 g/dL): number analyzed (Participants) | 21
  At Month 12 (>=10 g/dL) | 18
  At Month 12 (>=11 g/dL): number analyzed (Participants) | 21
  At Month 12 (>=11 g/dL) | 14
  At Month 12 (>=12 g/dL): number analyzed (Participants) | 21
  At Month 12 (>=12 g/dL) | 10
  At Month 12 (>=13 g/dL): number analyzed (Participants) | 21
  At Month 12 (>=13 g/dL) | 1
  At Month 12 (>=14 g/dL): number analyzed (Participants) | 21
  At Month 12 (>=14 g/dL) | 0
  At Month 18 (>=10 g/dL): number analyzed (Participants) | 19
  At Month 18 (>=10 g/dL) | 18
  At Month 18 (>=11 g/dL): number analyzed (Participants) | 19
  At Month 18 (>=11 g/dL) | 15
  At Month 18 (>=12 g/dL): number analyzed (Participants) | 19
  At Month 18 (>=12 g/dL) | 8
  At Month 18 (>=13 g/dL): number analyzed (Participants) | 19
  At Month 18 (>=13 g/dL) | 4
  At Month 18 (>=14 g/dL): number analyzed (Participants) | 19
  At Month 18 (>=14 g/dL) | 0
  At Month 24 (>=10 g/dL): number analyzed (Participants) | 20
  At Month 24 (>=10 g/dL) | 18
  At Month 24 (>=11 g/dL): number analyzed (Participants) | 20
  At Month 24 (>=11 g/dL) | 14
  At Month 24 (>=12 g/dL): number analyzed (Participants) | 20
  At Month 24 (>=12 g/dL) | 10
  At Month 24 (>=13 g/dL): number analyzed (Participants) | 20
  At Month 24 (>=13 g/dL) | 5
  At Month 24 (>=14 g/dL): number analyzed (Participants) | 20
  At Month 24 (>=14 g/dL) | 0

14. Secondary Outcome: Percentage of Participants Who Have Not Received Chelation Therapy for At Least 6 Months Following Drug Product Infusion
Description: Percentage of participants who have not received chelation therapy for at least 6 months following drug product infusion were reported.
Time Frame: Up to Month 24
Population: TP included all participants who received beti-cel.
Measure: Number; unit: percentage of participants
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 23
percentage of participants | 43.5

15. Secondary Outcome: Time From Last Iron Chelation Use to Last Follow-up
Description: Time from last iron chelation use to last follow-up to 24 months was reported. Participants were evaluable for this outcome if they had not received iron chelation therapy for at least 6 months following drug product infusion.
Time Frame: Time from last iron chelation up to Month 24 (actual maximum time frame of up to approximately 27 months due to visit window)
Population: TP population. Here, "Overall number of participants analyzed" signifies those participants who have not received chelation therapy for at least 6 months following drug product infusion. Data are presented through the Month 24 Visit based on calendar dates and including visit windows. Notably due to institutional COVID-19 restrictions and scheduling conflicts one participant had a Month 24 visit 42 days out of this window.
Measure: Median (Full Range); unit: months
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 10
months | 23.56 [17.6 to 24.6]

16. Secondary Outcome: Percentage of Participants Who Used Therapeutic Phlebotomy Post Drug Product (DP) Infusion
Description: Therapeutic phlebotomy could be used in lieu of chelation in participants who had Hb consistently >= 11 g/dL and who were no longer receiving regular transfusions, at the discretion of the investigator. Percentage of participants who used therapeutic phlebotomy post DP infusion for up to Month 24 were reported.
Time Frame: Up to Month 24
Population: TP included all participants who received beti-cel.
Measure: Number; unit: percentage of participants
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 23
percentage of participants | 30.4

17. Secondary Outcome: Annualized Phlebotomy Therapy Usage Following Drug Product Infusion
Description: Annualized phlebotomy therapy usage (number of procedures per year, calculated from DP infusion through last follow-up) were reported.
Time Frame: Up to Month 24
Population: TP included all participants who received beti-cel. Here, "Overall number of participants analyzed" signifies those participants who received therapeutic phlebotomy.
Measure: Mean (Standard Deviation); unit: number of procedures per year
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 7
number of procedures per year | 6.29 (4.786)

18. Secondary Outcome: Change From Baseline in Liver Iron Concentration by Magnetic Resonance Imaging (MRI)
Description: Change From Baseline in liver Iron Content by Magnetic Resonance Imaging (MRI) at Months 12 and 24 were reported.
Time Frame: Baseline, Months 12 and 24
Population: TP included all participants who received beti-cel. Participants were evaluable for this outcome if they had available liver iron content measurements at baseline and at the applicable follow-up timepoints. Here, "number of participants analyzed" signifies those participants who had LIC data available at Baseline, Months 12 and 24.
Measure: Mean (Standard Deviation); unit: milligrams per gram (mg/g)
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 22
milligrams per gram (mg/g)
  At Month 12 | 2.490 (4.1546)
  At Month 24 | 0.494 (3.9957)

19. Secondary Outcome: Change From Baseline in Cardiac T2* on MRI
Description: Change From Baseline in Cardiac T2* on MRI at baseline, Month 12 and 24 was reported.
Time Frame: Baseline, Months 12 and 24
Population: TP included all participants who received beti-cel. Participants were evaluable for this outcome if they had available cardiac T2* measurements at baseline and at the applicable follow-up timepoints. Here, "Overall number of participants analyzed" signifies those participants who had Cardiac T2* data available at Baseline, Months 12 and 24 and "number analyzed" signifies those participants at specific timepoint.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 21
milliseconds
  At Month 12: number analyzed (Participants) | 19
  At Month 12 | -1.0 (5.93)
  At Month 24 | -1.6 (7.42)

20. Secondary Outcome: Change From Baseline in Serum Ferritin at Months 12 and 24
Description: Serum ferritin was commonly used for an indirect estimation of body iron stores. Although sensitive, it is not specific for iron overload as it can be elevated in a variety of infectious and inflammatory states, and in the presence of cytolysis. Change from baseline in serum ferritin at Months 12 and 24 was reported.
Time Frame: Baseline, Months 12 and 24
Population: TP included all participants who received beti-cel. Participants were evaluable for this endpoint if they had available serum ferritin measurements at baseline and at the applicable follow-up timepoints. Here, "number analyzed" signifies those participants who were evaluable at specific timepoint.
Measure: Mean (Standard Deviation); unit: picomole per Liter (pmol/L)
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 23
picomole per Liter (pmol/L)
  At Month 12: number analyzed (Participants) | 22
  At Month 12 | 167.3 (1887.67)
  At Month 24 | -1163.8 (2435.58)

21. Secondary Outcome: Change From Baseline in Pediatric Quality of Life Inventory (PedsQL) Total Scores at Months 12 and 24
Description: PedsQL GCS designed to measure health-related quality of life in pediatric and adolescents (2 to 18 years). It encompassed 4 dimensions of functioning (physical [8 items], emotional [5 items], social [5 items], school [3 items]). Age groups: Toddler (2-4 years), Young pediatric (5-7 years), Pediatric (8-12 years), Teens (13-18 years). The questionnaire was also completed by parent/caregiver to assess parents' perceptions of their children's quality of life. The Toddler group consisted of 21 items, using a 5-point Likert scale (0 to 4); all other groups consisted of 23 items, with a 3-point Likert scale (0, 2, 4) for young pediatric, a 5-point Likert scale for pediatric and teens groups. All reported scores were transformed on a scale from 0 to 100 for each domain where 0=100, 1=75, 2=50, 3=25, and 4=0. Higher scores correspond with higher quality of life.
Time Frame: Baseline, Months 12 and 24
Population: TP included all participants who received beti-cel. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were <18 years at specific timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 14
Score on a scale
  Parent total score: Change at Month 12: number analyzed (Participants) | 12
  Parent total score: Change at Month 12 | 8.76 (12.071)
  Parent total score: Change at Month 24 | 6.03 (9.753)
  Patient total score: Change at Month 12: number analyzed (Participants) | 11
  Patient total score: Change at Month 12 | 6.82 (16.079)
  Patient total score: Change at Month 24: number analyzed (Participants) | 12
  Patient total score: Change at Month 24 | 9.96 (16.997)

22. Secondary Outcome: Change From Baseline in EuroQol Quality of Life 5-Dimension Youth Scale (EQ-5D-Y) VAS Health Status at Months 12 and 24
Description: EQ-5D is a validated, standardized, generic instrument that was most widely used preference based health related quality of life questionnaire in cost effectiveness and health technologies assessment. EQ-5D-Y was a version of instrument specifically developed and validated for use by youths aged 12 through 17 years. The EQ-5D-Y visual analog scale (VAS) consisted of a 20-cm vertical VAS, with anchors of 0 ("worst imaginable health state") and 100 ("best imaginable health state"). Respondents were asked to rate their own health state today by drawing a line from a box containing these words to the point on the scale that they felt most accurately reflected their current health state. The VAS was reported (raw data) on a scale of 0-100 where 0= death and 100= perfect health. Higher scores equated to better outcomes.
Time Frame: Baseline, Months 12 and 24
Population: TP included all participants who received beti-cel. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were 11 to <18 years at specific timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 7
Score on a scale
  Health State: Change at Month 12: number analyzed (Participants) | 6
  Health State: Change at Month 12 | 15.8 (20.60)
  Health State: Change at Month 24 | 20.9 (18.86)

23. Secondary Outcome: Change From Baseline in EuroQol Quality of Life 5-Dimension Adult Scale (EQ-5D-3L) VAS Heath Status Score at Months 12 and 24
Description: EQ-5D is a validated, standardized, generic instrument that was most widely used preference based health related quality of life (HRQoL) questionnaire in cost effectiveness and health technologies assessment. Participants age >=18 at time of informed consent were eligible to complete the EQ-5D-3L which is a visual analog scale (VAS) which consists of a 20-cm vertical VAS, with anchors of 0 ("worst imaginable health state") and 100 ("best imaginable health state"). Respondents were asked to rate their own health state today by drawing a line from a box containing these words to the point on the scale that they feel most accurately reflects their current health state.
Time Frame: Baseline, Months 12 and 24
Population: TP included all participants who received beti-cel. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this endpoint and number analyzed signifies those participants who were >= 18 years at specific timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 9
Score on a scale
  Health state: Change at Month 12 | 6.9 (11.93)
  Health state: Change at Month 24 | 9.7 (14.91)

24. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) Questionnaire Score
Description: FACT-BMT is assessed bone marrow transplant related quality of life in adults. It. Total score was sum of sub-scale scores for 5 domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, and Bone Marrow Transplantation Subscale. Each item scored on a 5-point Likert scale based on participant agreement with each statement: 0 for "not at all," 1 for "a little bit," 2 for "somewhat," 3 for "quite a bit," and 4 for "very much. Reported scores were transformed as follows: After taking into account reverse scores for questions constructed in negative form, subscale score for each domain was calculated by multiplying sum of item scores by number of items in subscale, then dividing by number of items answered. Total score was sum of subscale total added together and ranges from 0-148. Higher scores corresponded with higher quality of life.
Time Frame: Baseline, Months 12 and 24
Population: TP included all participants who received beti-cel. Here, "Overall number of participants analyzed" signifies those participants who were >= 18 years for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 9
Score on a scale
  Total Score: Change at Month 12 | 3.78 (16.994)
  Total Score: Change at Month 24 | 2.15 (13.695)

25. Secondary Outcome: Change From Baseline in Short Form-36 Health Survey (SF-36), Version 2, Acute (Physical and Mental Component Summary Scores) at Months 12 and 24
Description: SF-36 was designed to measure health-related quality of life in adults. The instrument consisted of 36 items, were aggregated into 8 multi-item scales (physical functioning [1=yes, limited a lot to 3=no, not limited at all], role-physical [1=all of time to 5=none of time], bodily pain [1=very severe to 6=none], general health [1=poor to 5=excellent], vitality [1=none of time to 5=all of time], social functioning [1=all of time: to 5=none of time], role emotional [1=all of time to 5=none of time] and mental health [1=all of time to 5=none of the time]). Four domains comprised physical component summary (PCS) score (physical functioning, role-physical, bodily pain, general health) and remaining 4 domains comprised mental component summary (MCS) score (vitality, social functioning, role-emotional, mental health). Reported summary scores were transformed on a scale from 0 to 100. Higher scores corresponded with higher quality of life.
Time Frame: Baseline, Months 12 and 24
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 9
Score on a scale
  Physical Component: Change at Month 12 | 0.80 (4.838)
  Physical Component: Change at Month 24 | 0.82 (3.672)
  Mental Component: Change at Month 12 | 1.88 (8.201)
  Mental Component: Change at Month 24 | 0.93 (10.805)

ADVERSE EVENTS:
Time Frame: From date of informed consent up to Month 24
Description: ITT population included all participants who initiated mobilization procedure.
Groups:
- LentiGlobin BB305 Drug Product: Participants aged <= 50 years received a single IV infusion of LentiGlobin BB305 Drug Product at a dose of >= 5.0 × 10^6 CD34+ cells/kg following myeloablative conditioning with busulfan (termed the Transplant population).
Arm/Group | LentiGlobin BB305 Drug Product
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 14/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LentiGlobin BB305 Drug Product (N=24)
Contusion (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1
Hypotension (Vascular disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Pyrexia (General disorders) | 3
Catheter site haemorrhage (General disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Venoocclusive liver disease (Hepatobiliary disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Neutropenic sepsis (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Device related sepsis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Vascular device infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LentiGlobin BB305 Drug Product (N=24)
Catheter site pain (General disorders) | 3
Chest pain (General disorders) | 4
Fatigue (General disorders) | 4
Mucosal inflammation (General disorders) | 3
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 3
Pyrexia (General disorders) | 12
Anxiety (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 3
Ligament sprain (Injury, poisoning and procedural complications) | 2
Procedural pain (Injury, poisoning and procedural complications) | 11
Skin abrasion (Injury, poisoning and procedural complications) | 2
Transfusion reaction (Injury, poisoning and procedural complications) | 3
Activated partial thromboplastin time prolonged (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 6
Blood alkaline phosphatase increased (Investigations) | 3
Blood magnesium decreased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 5
Palpitations (Cardiac disorders) | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 17
Febrile neutropenia (Blood and lymphatic system disorders) | 8
Leukocytosis (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 13
Lymphopenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 24
Headache (Nervous system disorders) | 10
Vertigo (Ear and labyrinth disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 9
Abdominal pain upper (Gastrointestinal disorders) | 2
Anal fissure (Gastrointestinal disorders) | 2
Anal haemorrhage (Gastrointestinal disorders) | 3
Anal inflammation (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 4
Gingival bleeding (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 14
Stomatitis (Gastrointestinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 16
Haematuria (Renal and urinary disorders) | 3
Venoocclusive liver disease (Hepatobiliary disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 8
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 5
Fluid overload (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 4
Cellulitis (Infections and infestations) | 2
Folliculitis (Infections and infestations) | 4
Gingivitis (Infections and infestations) | 2
Molluscum contagiosum (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 3
Rhinitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/02/NCT02906202/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/02/NCT02906202/SAP_001.pdf